CLINICAL TRIAL: NCT03774745
Title: A Randomized Trial of Mifepristone Antagonization With High-Dose Progesterone to Prevent Medical Abortion
Brief Title: Blocking Mifepristone Action With Progesterone
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Safety
Sponsor: University of California, Davis (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1353650
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy, Unwanted
Keywords: mifepristone; progesterone; abortion
MeSH Terms: interventions — Mifepristone; Progesterone

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo pills in opaque bottle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Progesterone (Experimental): Micronized progesterone 200mg oral capsules starting 24 hours after mifepristone 200mg ingestion (day 1).
  Progesterone treatment days 2-4: two capsules twice daily orally. Progesterone treatment days 5-15, 16 or 17: two capsules once daily orally.
  Interventions: Drug: Mifepristone 200 MG; Drug: micronized Progesterone
- Placebo oral capsule (Placebo Comparator): Placebo capsules starting 24 hours after mifepristone 200mg ingestion (day 1). Placebo treatment days 2-4: two capsules twice daily orally. Placebo treatment days 5-15, 16 or 17: two capsules once daily orally.
  Interventions: Drug: Mifepristone 200 MG; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Mifepristone 200 MG — All subjects receive mifepristone tablet on treatment day 1.
  Other Names: Mifeprex
Drug: micronized Progesterone — Subjects randomized to progesterone receive treatment starting day 2.
  Other Names: Prometrium
  Arms: Progesterone
Drug: Placebo oral capsule — Subjects randomized to placebo receive treatment starting day 2.
  Other Names: Placebo (for micronized progesterone)
  Arms: Placebo oral capsule

SUMMARY:
Double-blind randomized trial to evaluate the potential impact of progesterone treatment on early pregnancies exposed to mifepristone.

DETAILED DESCRIPTION:
Medical abortion commonly refers to early pregnancy termination (usually before 10 weeks' gestation) performed without primary surgical intervention and resulting from the use of abortion-inducing medications. The use of medications to cause abortion has been around for almost 70 years but the modern era of medical abortion treatment evolved with the development of mifepristone, a progesterone-receptor blocker with an affinity for the receptor greater than progesterone itself.

Medical abortion with mifepristone and misoprostol is highly effective; however, the risk of continuing pregnancy is still present, especially as gestation advances. While most women opt for further treatment in these scenarios, such as surgical aspiration, there are some who decide to continue the pregnancy. Thus, even following treatment, some women do change their mind.

No well-done study has evaluated whether such treatment works. Poorly controlled case series are not evidence and systematic reviews of continuing pregnancy rates after mifepristone/prostaglandin analogue treatment failure do not reflect real life outcomes. This study is also a first step to understanding if large studies evaluating mifepristone antagonization with high-dose progesterone are indicated and if placebo-controlled randomized trials can be successfully completed when evaluating this question.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant females 18 years and older at enrollment.
2. Seeking surgical abortion at 44-63 days' gestation on Study day 1.
3. Have received counseling and signed informed consent per UCD standard procedures for surgical abortion.
4. Presence of embryonic gestational cardiac activity on transvaginal ultrasonography.
5. English-speaking
6. Willing to sign informed consent and follow study protocol.
7. Willing to experience potential expulsion of the pregnancy with mifepristone treatment.

Exclusion Criteria:

1. Medical contraindications to medical abortion.

   1. Poorly controlled hypertension (systolic BP >160 or diastolic BP >95)
   2. Significant anemia - known recent hemoglobin <9.5 gm/dL
   3. Clinically significant cardiovascular disease (angina, valvular disease, arrhythmia, or congestive heart failure)
   4. Breastfeeding
   5. Coagulopathy or therapeutic coagulation
   6. Ultrasound evidence of molar or ectopic pregnancy
   7. Chronic systemic corticosteroid use
   8. Adrenal disease
   9. Sickle cell anemia with frequent/recent crises
   10. Glaucoma
2. IUD in place during conception, even if removed.
3. Peanut allergy.
4. Known intolerance of mifepristone or progesterone.
5. Any other condition, that in the opinion of the clinician, would contraindicate mifepristone, progesterone or medical abortion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologic females who are pregnant
Enrollment: 12 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Creinin, MD, Principal Investigator — University of California, Davis
Locations (3):
- United States (3):
  - Planned Parenthood Mar Monte, Sacramento, California
  - University of California, Davis, Sacramento, California
  - Family Planning Associates, Sacramento, California

IPD SHARING:
Plan to Share IPD: No
Sharing de-identified data will be considered upon individual request

REFERENCES:
- [Derived] Creinin MD, Hou MY, Dalton L, Steward R, Chen MJ. Mifepristone Antagonization With Progesterone to Prevent Medical Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jan;135(1):158-165. doi: 10.1097/AOG.0000000000003620. PMID 31809439

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone: Micronized progesterone 200mg oral capsules starting 24 hours after mifepristone 200mg ingestion (day 1).
  Progesterone treatment days 2-4: two capsules twice daily orally. Progesterone treatment days 5-15, 16 or 17: two capsules once daily orally.
  Mifepristone 200 MG: All subjects receive mifepristone tablet on treatment day 1.
  micronized Progesterone: Subjects randomized to progesterone receive treatment starting day 2.
Period: Overall Study
Arm/Group | Progesterone | Placebo Oral Capsule
Started | 6 | 6
Follow-Up 1 (3 +/- 1 day after enrollment) | 5 | 6
Follow-up 2 (7 +/1 day after enrollment) | 4 | 2
Completed (15 +/- 1 day after enrollment) | 4 | 2
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: Intended to enroll 40 total - study stopped after 12 enrolled due to safety concerns
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone | Placebo Oral Capsule | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 29.8 [24.6 to 39.6] | 24.1 [20.9 to 33.8] | 27.3 [20.9 to 39.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12
Gestational Age [Median (Full Range); unit: days] | 49.5 [47 to 56] | 55 [48 to 61] | 52.5 [47 to 61]
BMI [Median (Full Range); unit: kg/m^2] | 24.8 [19.0 to 36.4] | 24.6 [22.7 to 52.3] | 24.6 [19.0 to 52.3]
Obesity [Count of Participants; unit: Participants] | 2 | 2 | 4
Gravidity [Median (Full Range); unit: number of pregnancies] | 4.5 [1 to 10] | 3.5 [1 to 12] | 4 [1 to 12]
Parity [Median (Full Range); unit: number of deliveries] | 1.5 [0 to 6] | 0.5 [0 to 3] | 1 [0 to 6]
Past mifepristone use [Count of Participants; unit: Participants] | 1 | 3 | 4
Prior progesterone use (n, %) [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Continuing Pregnancy Based on Ultrasound Examination
Description: Pregnancy still in uterus with normal growth and gestational cardiac activity present based on ultrasound examination
Time Frame: at 14-16 days after mifepristone administration
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone | Placebo Oral Capsule
Number analyzed (Participants) | 6 | 6
Participants | 4 | 2

2. Secondary Outcome: Expulsion During Follow-up Evaluation
Description: Pregnancy expulsion following mifepristone treatment
Time Frame: up to 16 days after mifepristone administration
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone | Placebo Oral Capsule
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

3. Secondary Outcome: Number of Participants With Adverse Events During Follow-up Evaluation
Description: Side effects from progesterone/placebo treatment and ability to continued treatment as prescribed
Time Frame: up to 16 days after mifepristone administration
Population: increased to severe at any time during follow-up
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo Oral Capsule
Number analyzed (Participants) | 6 | 6
participants
  Nausea | 2 | 1
  Vomiting | 2 | 0
  Mastalgia | 0 | 0
  Tiredness | 0 | 1
  Mood changes | 1 | 0
  Reflux | 0 | 0
  Dizziness | 0 | 0
  Bleeding | 1 | 3
  Spotting | 0 | 0
  Cramping | 0 | 0

4. Secondary Outcome: Medical Safety During Treatment and Follow-up
Description: Adverse events related to morbidity, e.g. hemorrhage, emergency department visits, emergent dilation and curettage procedures
Time Frame: up to 16 days after mifepristone administration
Population: intent to treat
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo Oral Capsule
Number analyzed (Participants) | 6 | 6
participants
  Hemorrhage | 1 | 2
  Emergency Room Visit | 1 | 2
  Transfusion | 0 | 1
  Emergent D&C | 0 | 2
  Side effects - request D&C | 1 | 1

5. Secondary Outcome: Number of Participants With Change in Serum Progesterone and hCG During Follow-up
Description: Change in serum progesterone and hCG during follow-up evaluation
Time Frame: up to 16 days after mifepristone administration
Population: intent to treat
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo Oral Capsule
Number analyzed (Participants) | 6 | 6
participants
  Progesterone increase from baseline at FU 1 | 5 | 2
  Progesterone decrease from baseline at FU 1 | 0 | 2
  hCG increase from baseline at FU 1 | 4 | 3
  hCG decrease from baseline at FU 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: Two weeks
Description: Adverse event included hemorrhage, emergency room visit, transfusion, emergent D&C
Arm/Group | Progesterone | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=6) | Placebo Oral Capsule (N=6)
Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Transfusion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Emergency D&C (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Emergency Room Visit (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=6) | Placebo Oral Capsule (N=6)
Side effects requesting study discontinuation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Requested D&C for abortion because could not tolerate medications/pregnancy

LIMITATIONS AND CAVEATS:
Early termination for safety reasons leading to small numbers of subjects analyzed for efficacy outcomes. Imbalance in participant characteristics due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03774745/Prot_SAP_000.pdf